CLINICAL TRIAL: NCT01166516
Title: A Prospective Study With the IBV Valve System for the Treatment of Prolonged Air Leak
Brief Title: IBV Valve System for the Treatment of Prolonged Air Leak Under HDE H060002 - Post Approval Study
Acronym: HUD-PAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Olympus Corporation of the Americas (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPR-02704
Record Dates: First submitted 2010-07-13; First posted 2010-07-21 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Prolonged Air Leak
Keywords: Prolonged air leak; lobectomy; segmentectomy; lung volume reduction surgery (LVRS)
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment with HUD IBV Valve System (Other): Treatment with HUD IBV Valve System in Post-Approval Study
  Interventions: Device: Treatment with HUD IBV Valve System

INTERVENTIONS:
Device: Treatment with HUD IBV Valve System — Treatment involves placing one or more valves in the airways of the lung to control a prolonged air leak.
  Other Names: IBV Valve System

SUMMARY:
Study to collect post-market safety data for HUD IBV Valve System, a device to control prolonged air leaks of the lung, or significant air leaks that are likely to become prolonged air leaks following lobectomy, segmentectomy, or LVRS. An air leak present on post-operative day 7 is considered prolonged unless present only during forced exhalation or cough. An air leak present on day 5 should be considered for treatment if it is: 1)continuous, 2) present during normal inhalation phase of inspiration, or 3) present upon normal expiration and accompanied by subcutaneous emphysema or respiratory compromise.

ELIGIBILITY:
Inclusion Criteria:

* Subject has an air leak present on day 7 after lobectomy, segmentectomy, or lung volume reduction surgery (LVRS), or on day 5 if the air leak is 1) continuous, 2) present during normal inhalation phase of inspiration, or 3) present upon normal expiration and accompanied by subcutaneous emphysema or respiratory compromise

Exclusion Criteria:

* Air leak only on force exhalation or cough
* Subject has significant active asthma, pneumonia, bacterial bronchitis or clinically significant bronchiectasis
* Subject is unable to provide informed consent and there is no designated authority to sign for the incapacitated patient
* Subject is not an appropriate candidate for, or unable to tolerate, flexible bronchoscopy procedures
* Subject has co-morbidities or factors that will prevent follow-up during the study period

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-04; Primary Completion 2016-03 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Safety | Day 0 to 6 weeks
  The primary objective of this study is to characterize the device safety profile. Adverse events (AEs) reported during the study will be analyzed and summarized. This information will be used to enhance the HDE device labeling.

SECONDARY OUTCOMES:
Probable Benefit | Day 0 to 6 weeks
  Secondary study objectives are to gather probable benefit information regarding reduction in air leaks and reduction in health care utilization to support potential future premarket applications. The response of the air leak to valve treatment will be observed and recorded along with the time of observation. Probable benefit information gathered during the study will be analyzed and summarized

CONTACTS AND LOCATIONS:
Overall Officials: Douglas E. Wood, MD, Principal Investigator — University of Washington
Locations (13):
- United States (13):
  - Piedmont Hospital, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - SIU School of Medicine, Springfield, Illinois
  - Olathe Medical Center, Olathe, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Lahey Clinic, Burlington, Massachusetts
  - Cleveland Clinic, Cleveland, Ohio
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - UT Southwestern Medical Center at Dallas, Dallas, Texas
  - Michael DeBakey VA Medical Center, Houston, Texas
  - Swedish Medical Center, Seattle, Washington
  - University of Washington, Seattle, Washington